CLINICAL TRIAL: NCT03624283
Title: The Effect of Vestibular Exercise, With or Without Medication, in Managing Residual Dizziness After Successful Repositioning Maneuvers in Patients With Benign Paroxysmal Positional Vertigo
Brief Title: Interventions for Residual Dizziness After Successful Repositioning Maneuvers in Patients With BPPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Huawei Li, Ph.D, MD, Director of Otorhinolaryngology, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vestibular rehabilitation
Record Dates: First submitted 2018-07-31; First posted 2018-08-10 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases | interventions — Betahistine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A will be provided with Exercise-based vestibular rehabilitation (VR) twice per day for a period of 4 weeks;
  Interventions: Behavioral: Exercise-based vestibular rehabilitation
- Group B (Experimental): Group B will be prescribed with Betahistine 12mg, twice daily for 7 days;
  Interventions: Drug: Betahistine
- Group C (Experimental): Group C will receive an combination of Exercise-based VR plus Betahistine.
  Interventions: Drug: Betahistine; Behavioral: Exercise-based vestibular rehabilitation

INTERVENTIONS:
Drug: Betahistine — Betahistine is used in the treatment of and vertigo.
  Arms: Group B; Group C
Behavioral: Exercise-based vestibular rehabilitation — Exercise-based vestibular rehabilitation (VR) has proven to be an effective way for managing dizziness by relieving symptoms and improving balance and postural stability.
  Arms: Group A; Group C

SUMMARY:
To investigate the effect of vestibular rehabilitation, with or without medication, on resolving residual dizziness after successful repositioning maneuvers in patients with benign paroxysmal positional.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as unilateral BPPV (unilateral posterior semicircular canal BPPV or horizontal semicircular canal BPPV) according to the clinical practice guideline issued by American Academy of Otolaryngology and head and neck surgery (AAO-HNSF) in 2017;
2. Aged 18~80 years;
3. Reporting residual symptoms after successful repositioning maneuvers;

Exclusion Criteria:

1. Anterior semicircular canal BPPV or multicanal BPPV;
2. Recurrent BPPV;
3. Subjects with coexisting vestibular disorders, including Meniere disease, vestibular neuritis, labyrinthitis, and peripheral vestibular loss;
4. Subjects with severe cervical spine disease;
5. Subjects with severe cardiovascular diseases ;
6. Subjects with known cerebral vascular disease like carotid stenosis;
7. Cognitive impairment;
8. Suspect of significant depression or anxiety as defined as a score of ≥ 8 for each respective scale of Hospital anxiety and depression scale;
9. Pregnant/ lactating or planning to become pregnant during the study period;
10. Had taken vestibulosupressant, antihistamines, and/ or ototoxic medications in the past 3 months;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Balance function | Change from baseline, at 4 weeks, 8 weeks and 12 weeks postrandomisation
  Balance function, measured by computerized dynamic posturography.

SECONDARY OUTCOMES:
Duration of RD symptoms | Change from baseline at 4 weeks, 8 weeks and 12 weeks postrandomisation.
  Patients self-reported days for RD onset to disappear
Quality of life assessment scale | Change from baseline at 4 weeks, 8 weeks and 12 weeks postrandomisation.
  Measured by Dizziness and Handicap Inventory
Otolith function | Change from baseline at 4 weeks, 8 weeks and 12 weeks follow-up will be necessary only when the previous examine showing abnormal.
  Analyzed as vestibular evoked myogenic potenials (VEMPs)
Daily function | Change from baseline, at 4 weeks, 8 weeks and 12 weeks postrandomisation
  Daily function quantified by Vestibular Activities and Participation (VAP) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu P, Cao W, Hu Y, Li H. Effects of vestibular rehabilitation, with or without betahistine, on managing residual dizziness after successful repositioning manoeuvres in patients with benign paroxysmal positional vertigo: a protocol for a randomised controlled trial. BMJ Open. 2019 Jun 18;9(6):e026711. doi: 10.1136/bmjopen-2018-026711. PMID 31217316